CLINICAL TRIAL: NCT05804682
Title: Fascial Versus Standard Neck Dissection in Patients With N1b Papillary Thyroid Carcinoma: a 4-year Analysis of Outcomes.
Brief Title: Fascial Versus Standard Neck Dissection in Patients With N1b Papillary Thyroid Carcinoma
Acronym: FADO
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4818
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2022-03

CONDITIONS: Patients With Papillary Thyroid Cancer and N1b Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients that underwent fascial dissection for N1b papillary thyroid cancer
  Interventions: Procedure: Fascial Neck Dissection
- Patients that underwent ftandard dissection for N1b papillary thyroid cancer
  Interventions: Procedure: Standard Neck Dissection

INTERVENTIONS:
Procedure: Fascial Neck Dissection — Central and lateral neck dissection with the fascial technique
  Groups: Patients that underwent fascial dissection for N1b papillary thyroid cancer
Procedure: Standard Neck Dissection — Central and lateral neck dissection with the standard technique
  Groups: Patients that underwent ftandard dissection for N1b papillary thyroid cancer

SUMMARY:
Optimal surgical technique for neck dissection (LND) in thyroid carcinoma remains a subject of debate. Fascial ND (FND) implies the removal of the superficial and middle layers of the deep cervical fascia en bloc with lymph-nodes containing fibro-fatty tissue (levels IIa-Vb and VI-VII for cN1b patients). This retrospective cohort study was designed to compare FND with standard, non-fascial, selective ND (SND).

DETAILED DESCRIPTION:
In thyroid cancer patients, lymph node dissection includes a comprehensive removal of all the target nodal basins: anterior cervical compartment (level VI) and the superior mediastinal nodes that can be reached via cervical incision (level VII) in CND, and levels IIa-Vb in LND. Clearance of those levels without including the enveloping fasciae in the specimen is referred to hereafter as Standard Neck Dissection (SND), as it is the most common technique applied for thyroid tumors. In Fascial Neck Dissection, the comprehensive clearance of the target basins is achieved by following the planes of coalescence of the cervical fascial layers. Those are avascular and enable the removal of the target nodes en bloc with their investing fascial layers.

The aim of this retrospective study was to compare the outcomes between fascial and standard approach in N1b PTC patients that underwent surgery for N1b papillary thyroid cancer. The primary objective was to achieve a significantly higher nodal yield by applying the fascial neck dissection technique and reduce rates of early loco-regional recurrence. Secondary objectives were the evaluation of short and long-term post-operative complications and the cosmetic result.

ELIGIBILITY:
Inclusion Criteria:

Patients who met all the following criteria were eligible for inclusion in this retrospective evaluation:

* Male or female patients, living or deceased, aged 18 years or older at the time of operation
* Unilateral (left/right) or bilateral lateral neck dissection along with central neck dissection
* Patients with papillary cancer, pN1b. This excludes patients with other types of thyroid cancer (e.g., medullary, follicular, and anaplastic);
* Patients that underwent central and/or lateral neck dissection as a primary intervention. This excludes patients with any previous operation for thyroid disease involving any type of lymph node dissection.

Exclusion criteria: patient's age < 18 years, patients that underwent previous neck dissection of any type and patients who refused or were unable to provide adequate follow up data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that were operated for N1b papillary thyroid cancer in the Division of Endocrine and Metabolic Surgery, Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy between 2018 and 2021. All patients eligible for inclusion were screened for eligibility in a systematic fashion both from the records of our center in the Eurocrine registry and from our center's internal prospective de-identified database concerning thyroid cancer.
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Early loco-regional recurrence | Interventions 2018-2021, Final follow up January 2023
  Locoregional recurrence within 1 year from operation
Harvested lymph nodes | Interventions 2018-2021, Final follow up January 2023
  Total and positive lymph node yields for central and lateral compartments

SECONDARY OUTCOMES:
Early and late complications | Interventions 2018-2021, Final follow up January 2023
Voice and swallowing score comparisons | Interventions 2018-2021, Final follow up January 2023
Cosmetic outcome | Interventions 2018-2021, Final follow up January 2023

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Only after individual contact by researchers of the field